CLINICAL TRIAL: NCT02694731
Title: A Mindfulness Mobile Intervention Targeting Reductions in Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-17250
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Food Cravings
Keywords: Craving; Mobile Apps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile application intervention (Experimental): Participants receive a mobile app with a 5-week mindful eating program and ongoing tools for coping with cravings
  Interventions: Behavioral: Mobile application intervention (Device: Smartphone)

INTERVENTIONS:
Behavioral: Mobile application intervention (Device: Smartphone) — Consists of the app described in the arm description.

SUMMARY:
Participants will complete a 5-week smartphone app-based intervention that teaches mindful eating skills. One goal is to determine to what extent participants will enjoy using the app and complete the intervention. The investigators predict that after completing the intervention, participants will report fewer episodes of eating in response to food cravings. The investigators will also measure several other biological and behavioral outcomes.

DETAILED DESCRIPTION:
In this prospective repeated-measures cohort study, participants will complete a 5-week smartphone app-based intervention that teaches mindful eating skills. The investigators will assess psychological and behavioral intervention targets using questionnaires and brief mobile assessments. The investigators will also measure BMI and adiposity. Assessments will occur at pre-intervention, post-intervention, and 1 and 2 months post intervention. At several times during the study, participants will also receive multiple daily text messages asking them to complete a brief food craving assessment on their phone. This "experience sampling" approach is critical as it allow the investigators to capture experiences and behaviors that are often brief and automatic, making them poorly suited to traditional retrospective questionnaires. The investigators will also assess acceptability and continued use of the app via anonymous usage logs.

Overall, the aims are to 1) assess feasibility of the protocol, 2) assess changes in food cravings and indulgence of cravings, and 3) determine the extent to which participants remain engaged with the app after completing the 5-week intervention period and whether this predicts maintenance of benefits at 1 month and 2 months post-intervention. An exploratory aim is to measure the effects of the intervention on body weight, bodyfat, and bodyfat distribution.

ELIGIBILITY:
Inclusion Criteria:

* Problems with controlling food intake as indexed by "yes" responses to the following two questions: "Do you have food cravings?" and "Do you eat in response to your food cravings more than you would like to?"
* Overweight or obese (BMI of 25.0 to 39.9 kg/m2)
* Score at or above the scale midpoint on the Readiness Ruler, a single-item visual analog scale measure of readiness for behavioral change (prompt is, "I have decided to give in to food cravings less")
* Have and use a smartphone (Android or iOS) with internet access.
* Report food cravings on most days and a desire to indulge in food cravings less

Exclusion Criteria:

* Current diabetes
* Pregnant or plans to become pregnant within 4 months
* Current diagnosis of anorexia or bulimia
* In the opinion of an investigator, meets any of the following criteria:

  1. Likely to drop out due to expressed ambivalence or lack of interest
  2. Likely to be harmed in any way by participating
  3. Likely to have provided untruthful answers to the screening questions (based on evidence such as unclear or inconsistent responses when talking to study staff vs. reporting online, or log data showing repeated attempts to "game" the screening questionnaire).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Craving indulgence frequency | 1 month post-intervention
  Cell phone questionnaires assess frequency with which participants eat in response to food cravings. Cell phone questionnaires assess frequency with which participants eat in response to food cravings. Participants are asked whether they ate in response to a craving in the past hour

SECONDARY OUTCOMES:
Craving indulgence frequency | Administered 9 times over the 7 days after the participant completes the intervention (typically 28 days after beginning the study; may be longer if participant takes extra days to complete the intervention)
  Cell phone questionnaires assess frequency with which participants eat in response to food cravings. Participants are asked whether they ate in response to a craving in the past hour
Reward-based Eating Drive (RED) | 1 month post-intervention
  Questionnaire measure of drive to eat for hedonic properties of food
Reward-based Eating Drive (RED) | immediate post-intervention (within 7 days of completing the intervention)
  Questionnaire measure of drive to eat for hedonic properties of food
Palatable Eating Motives Scale, coping subscale | 1 month post-intervention
  Questionnaire measure of drive to eat for coping
Palatable Eating Motives Scale, coping subscale | Immediate post-intervention (within 7 days of completing the intervention)
  Questionnaire measure of drive to eat for coping
Food Cravings Questionnaire (FCQ-T-R) | 1 month post-intervention
  Questionnaire measure of food cravings
Food Cravings Questionnaire (FCQ-T-R) | Immediate post-intervention (within 7 days of completing the intervention)
  Questionnaire measure of food cravings

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will deposit anonymized individual-level data in a depository such as the Open Science Framework.

REFERENCES:
- [Background] Wansink B. Environmental factors that increase the food intake and consumption volume of unknowing consumers. Annu Rev Nutr. 2004;24:455-79. doi: 10.1146/annurev.nutr.24.012003.132140. PMID 15189128
- [Background] Gendall KA, Joyce PR, Sullivan PF. Impact of definition on prevalence of food cravings in a random sample of young women. Appetite. 1997 Feb;28(1):63-72. doi: 10.1006/appe.1996.0060. PMID 9134095
- [Background] Epel ES, Tomiyama AJ, Mason AE, Laraia BA, Hartman W, Ready K, Acree M, Adam TC, St Jeor S, Kessler D. The reward-based eating drive scale: a self-report index of reward-based eating. PLoS One. 2014 Jun 30;9(6):e101350. doi: 10.1371/journal.pone.0101350. eCollection 2014. PMID 24979216
- [Derived] Sagui-Henson SJ, Radin RM, Jhaveri K, Brewer JA, Cohn M, Hartogensis W, Mason AE. Negative Mood and Food Craving Strength Among Women with Overweight: Implications for Targeting Mechanisms Using a Mindful Eating Intervention. Mindfulness (N Y). 2021;12(12):2997-3010. doi: 10.1007/s12671-021-01760-z. Epub 2021 Sep 24. PMID 34584574
- [Derived] Mason AE, Jhaveri K, Cohn M, Brewer JA. Testing a mobile mindful eating intervention targeting craving-related eating: feasibility and proof of concept. J Behav Med. 2018 Apr;41(2):160-173. doi: 10.1007/s10865-017-9884-5. Epub 2017 Sep 16. PMID 28918456